CLINICAL TRIAL: NCT02766218
Title: Mealtime Interactions and Risk of Obesity in Toddlers
Brief Title: Mealtime Interactions and Risk of Toddler Obesity
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Collaborators: The Miriam Hospital (Other); California Polytechnic State University-San Luis Obispo (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23356; R01DK108661 (NIH); R56DK108661 (NIH)
Record Dates: First submitted 2016-02-12; First posted 2016-05-09 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obesity
Keywords: toddler obesity; responsive feeding; behavioral weight control; pregnancy weight gain; early life risk factors
MeSH Terms: conditions — Obesity; Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Behavioral: Lifestyle Intervention: The intervention is a multicomponent program designed to prevent excessive gestational weight gain in obese women through modifications of diet, exercise, and behavioral strategies during pregnancy.
- No Intervention: Standard Care

SUMMARY:
The purpose of this observational study is to conduct 18-, 24-, and 36-month assessments with mother-toddler dyads who participated in a study that is testing the effects of a multicomponent lifestyle intervention as a means to prevent excessive gestational weight gain in obese women. Specifically, dyads will be invited to participate in home-based assessments to videotape an evening meal, have anthropometric measures taken, and complete study questionnaires. The overall goal is to understand factors related prospectively to responsive feeding between mothers and toddlers at 18 months; determine whether responsive feeding at 18 and 24 months predicts change in zBMI and adiposity from 18-36 months; and explore which factors are most strongly predictive of child zBMI change from birth to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Mother participated in clinical trial #NCT01545934
* Child 18-36 months old

Exclusion Criteria:

* Child chronic health conditions that could affect feeding or growth (diagnosed feeding disorders, use of feeding tube) or could influence the mealtime interaction (significant food allergies or dietary restrictions, diagnosed psychiatric disorders, or pervasive developmental delays).

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Mothers and their 18-month-old toddlers who participated in clinical trial #NCT01545934 will be invited to participate in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Responsive feeding | 18- and 24-months
  The Responsiveness to Child Feeding Cues Scale will be used to code maternal responsive feeding. Primary outcomes are: a) maternal responsiveness to toddler fullness cues.

SECONDARY OUTCOMES:
Child Weight Status | birth, 6-, 12-, 18-, 24- and 36-months
  zBMI will be computed at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Chantelle Hart, PhD, Principal Investigator — Temple University; Suzanne Phelan, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo; Rena Wing, PhD, Principal Investigator — The Miriam Hospital

IPD SHARING:
Plan to Share IPD: No